CLINICAL TRIAL: NCT02953730
Title: The Study on the Pharmacokinetics of Pegylated Recombinant Human Granulocyte Stimulating Factor（PEG-rhG-CSF） in Children and Adolescents
Brief Title: The Study on the Pharmacokinetics of PEG-rhG-CSF in Children and Adolescents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Xiaofan Zhu, chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-JYL-05-01
Record Dates: First submitted 2016-11-01; First posted 2016-11-03 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Acute Lymphoid Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — pegylated granulocyte colony-stimulating factor

ARMS (1):
- PEG-rhG-CSF (Experimental)
  Interventions: Drug: PEG-rhG-CSF

INTERVENTIONS:
Drug: PEG-rhG-CSF

SUMMARY:
The purpose of the trail is to study the pharmacokinetics of Pegylated Recombinant Human Granulocyte Stimulating Factor（PEG-rhG-CSF） in Children and Adolescents

ELIGIBILITY:
Inclusion Criteria:

1. Age≤18 years old, gender no limited.
2. Patients with acute lymphoblastic leukemia diagnosed by bone marrow pathology or cytology.
3. Plan to receive CAM (cyclophosphamide,cytarabine,6-MP)chemotherapy regimen.
4. Previously not received radiotherapy.
5. Karnofsky Performance Scores ( KPS)≥60.
6. The expected survival time was >3 months.
7. Neutropenia or agranulocytosis, no bleeding tendency.
8. No significant cardiac dysfunction or metabolic disease.
9. TBIL(total bilirubin ), ALT（alanine aminotransferase）,AST（glutamic-oxalacetic transaminase） < 2.5×ULN（upper limit of normal）.
10. BUN（blood urine nitrogen），Cr（creatinine），UA（uric acid）<1.5×ULN.
11. Written informed consent are acquired.

Exclusion Criteria:

1. With a history of systemic radiotherapy.
2. Infection difficult to control, the body temperature ≥ 38℃.
3. Other situation that investigators consider as contra-indication for this study.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
peak concentration(Cmax) | 1 year
elimination half life(t 1/2kel) | 1 year
area under the curve(AUC) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofan Zhu, MD, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Department of Pediatrics, Institute of Hematology and Blood Disease Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China